CLINICAL TRIAL: NCT01763086
Title: Mesenchymal Stem Cells From Third-party Donors for Treatment of Poor Graft Function After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Mesenchymal Stem Cells for Treatment of Poor Graft Function After Allogeneic Hematopoietic Stem Cell Transplant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Sun Yat-sen University (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Southern Medical University, China (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFH-MSC-allo-HSCT-2013
Record Dates: First submitted 2013-01-05; First posted 2013-01-08 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Stem Cell Transplantation, Hematopoietic; Mesenchymal Stem Cells; Poor Graft Function; Hematological Diseases
Keywords: Poor Graft Function; Mesenchymal Stem Cells; Allogeneic hematopoietic stem cell transplantation; Third-party Donors
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stem cells (Experimental): Mesenchymal stem cells 1×10^6 cells/kg, intravenously
  Interventions: Biological: Mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells will be intravenously infused via a central venous catheter,at a dose of 1×10^6 cells/kg, over 15 min. The vital signs of all patients will be closely monitored during and for 24h after MSCs administration. If the NEU and PLT levels do not attain the completely response(CR)standards within 14d, a second course of MSCs treatment will be given.

SUMMARY:
The purpose of this study is to evaluate the utility of treating patients experiencing poor graft function after allogeneic hematopoietic stem cell transplantation with ex-vivo-expanded BM-drived mesenchymal stem cells from third-party donors. Our first objective was to evaluate the effect of such treatment on poor graft function, and second object was to investigate the safety of such treatment.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation(allo-HSCT) can cure many hematologic diseases. Although good progress has been made in the prevention and treatment of side effects associated with transplantation, poor graft function (PGF) remains an important complication that occurs in 5-27% of patients, and is associated with considerable morbidity and mortality related to infections or hemorrhagic complications. Treatment of PGF usually involves the prescription of hematopoietic growth factors such as granulocyte colony-stimulating factor (G-CSF), or repeat transplantation, but these methods are associated with short-term effect and a significant risk of graft-versus-host disease（GVHD） development, respectively.

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs are evolving rapidly with goals of improving hematopoietic engraftment, preventing and treating graft-versus-host disease after allo-HSCT and so on. However, the efficacy of treatment of PGF that develops after allo-HSCT using expanded BM-derived MSCs from a third-party donor is rarely reported. If such treatment could be shown to be effective and safe, BM-derived MSCs could potentially be used as an universal donor material. This would have a major impact because the generation of donor-specific MSCs is time-consuming, costly, and often impractical if the clinical status of a patient is urgent.

In the present study, the investigators will prospectively evaluate the efficacy and safety of ex-vivo-expanded BM-derived MSCs from third-party donors in treating patients with PGF after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 14-65 years
* Poor graft function developing after allo-HSCT
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
hematopoietic recovery | 1 year
  Hematopoietic reconstitution post-transplantation is defined as reconstitution of both neutrophil and platelet numbers. Neutrophil reconstitution is defined as occurring on the first 3 consecutive days with an neutrophil(NEU)>0.5×10^9/L, and platelet (PLT) reconstitution is defined as the first >20×10^9/L for 3 consecutive days.

SECONDARY OUTCOMES:
infections, primary underlying disease relapse and any toxic side effects of MSCs treatment | 1 year
  Infections will be mainly focused within the first 100 days after MSCs treatment. Toxic side effects of treatment includes acute toxicity and late side effects. Acute toxicity principally involves the heart,live and kidney. Late toxic side effects involves principally the development of secondary tumors and relapse of the primary disease.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Sanchez-Guijo FM, Lopez-Villar O, Lopez-Anglada L, Villaron EM, Muntion S, Diez-Campelo M, Perez-Simon JA, San Miguel JF, Caballero D, del Canizo MC. Allogeneic mesenchymal stem cell therapy for refractory cytopenias after hematopoietic stem cell transplantation. Transfusion. 2012 May;52(5):1086-91. doi: 10.1111/j.1537-2995.2011.03400.x. Epub 2011 Oct 24. PMID 22023454
- [Background] Meuleman N, Tondreau T, Ahmad I, Kwan J, Crokaert F, Delforge A, Dorval C, Martiat P, Lewalle P, Lagneaux L, Bron D. Infusion of mesenchymal stromal cells can aid hematopoietic recovery following allogeneic hematopoietic stem cell myeloablative transplant: a pilot study. Stem Cells Dev. 2009 Nov;18(9):1247-52. doi: 10.1089/scd.2009.0029. PMID 19309241